CLINICAL TRIAL: NCT01186263
Title: Exploratory Study to Assess the Predictive Value of 99mTc-labeled Albumin Spheres for the Intrahepatic Distribution of 90Y SIR Spheres in Patients With Liver Metastases of Colorectal Tumors
Brief Title: Predictive Value of 99mTc- Albumin Spheres Before 90Y- SIR Therapy
Acronym: EXPLOSIVE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Magdeburg (Other)
Collaborators: Sirtex Medical (Industry)
Responsible Party: Principal Investigator, Jens Ricke, Prof. Dr., University of Magdeburg
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: RAD050; 2008-005609-21 (EudraCT Number)
Record Dates: First submitted 2010-07-23; First posted 2010-08-23 (Estimated); Last update posted 2014-09-04 (Estimated); Status verified 2014-09

CONDITIONS: Colorectal Cancer; Liver Metastases
Keywords: liver metastases; MAA; B20; SIR spheres; SPECT; intra-hepatic distribution
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 99mTc- labeled albumin macroaggregates (MAA) (Experimental): Diagnostic MAA- SPECT- imaging.
  Interventions: Drug: MAA for diagnostic SPECT imaging
- 99mTc- labeled albumin microspheres (B20) (Experimental): Diagnostic B20- SPECT- imaging.
  Interventions: Drug: Diagnostic B20- SPECT imaging.

INTERVENTIONS:
Drug: MAA for diagnostic SPECT imaging — Intraarterial application of 5ml containing 500.000 particles with an activity of 150MBq.
  Other Names: TechneScan Lyo MAA
  Arms: 99mTc- labeled albumin macroaggregates (MAA)
Drug: Diagnostic B20- SPECT imaging. — Intraarterial application of 5ml containing 150.000 particles with an activity of 150 MBq.
  Other Names: ROTOP HSA microspheres B20
  Arms: 99mTc- labeled albumin microspheres (B20)

SUMMARY:
The purpose of this study is to assess the predictive value of 99mTechnetium (Tc)- labeled albumin in macroaggregates (MAA) and in microspheres (B20) injected into the common hepatic artery for the distribution of 90Yttrium- Selective Internal Radiotherapy (SIRT)-spheres (SIR- spheres).

DETAILED DESCRIPTION:
Patients with metastases of colorectal tumors will be included into this study provided that they are scheduled for 90Y SIR spheres therapy for clinical reasons. Before 90Y SIR spheres therapy, patients will receive a diagnostic examination with injection of MAA (group A) or B20 (group B) into the common hepatic artery to rule out a relevant shunt volume to the lung or other extra-hepatic locations (e.g., stomach) as recommended by the manufacturer. After the diagnostic scan, therapy with SIR- spheres will be conducted in 2 separate sessions with selective injection of 90Y labeled SIR spheres into the right and left hepatic artery at two separate occasions (routine procedure at the University of Magdeburg, Germany). In addition, therapeutic sessions will include the selective injection of MAA or B20 into the right / left hepatic artery according to a predefined plan (either alone or as a mixture with the SIR spheres).The intra-hepatic distribution of 90Y labeled SIR spheres will be assessed using "Bremsstrahlen"- Single- Photon- Emission- Computed- Tomography (SPECT)- imaging, the distribution of MAA and B20 will be assessed using SPECT imaging.

ELIGIBILITY:
Inclusion Criteria:

* age: between 18 and 85 years
* if female, postmenopausal or surgically sterilized
* liver metastases of a colorectal tumor in both liver lobes
* scheduled for therapy with 90Y SIR spheres for clinical reasons
* life expectancy longer than 6 months
* willing and able to undergo all study procedures
* having voluntarily provided written and fully informed consent

Exclusion Criteria:

* presenting with a contraindication to 90Y SIR spheres therapy
* variants of the arterial hepatic blood supply which interfere with the objectives of this study (e.g., variants of Michel)
* women who are pregnant, lactating or who are of childbearing potential
* patients being clinically unstable
* uncooperative, in the investigator's opinion
* any contraindication to SIRT treatment
* any concomitant chemotherapy
* shunt to the lung >10%
* shunt to any extrahepatic organ (except the lung)
* having been previously enrolled in this study
* participating in another prospective clinical trial

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2010-07; Primary Completion 2011-07 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Percentage of liver volume for which the accumulation of SIR spheres was correctly predicted by the preceding Tc-99m MAA scintigraphy | Tc-99m MAA scan one day prior to radioembolisation; Bremsstahlen-Scan after SIR spheres therapy
  The percentage in liver volume for which the accumulation of SIR spheres during therapy was correctly predicted by Tc-99m MAA will be given by a blinded reader in categories by visual assessment (0-10%, >10-20%, >20-30%, …, >90-100%) (only patients who received Tc-99m MAA during evaluation.)

SECONDARY OUTCOMES:
Percentage of liver volume for which the accumulation of SIR spheres was correctly predicted by the preceding Tc-99m B20 scintigraphy | Tc-99m B20 scan one day prior to radioembolisation; Bremsstahlen-Scan after SIR spheres therapy
  The percentage in liver volume for which the accumulation of SIR spheres during therapy was correctly predicted by B20 will be given by a blinded reader in categories by visual assessment (0-10%, >10-20%, >20-30%, …, >90-100%) (only patients who received Tc-99m B20 during evaluation.)
Pharmacokinetic parameters of the intrahepatic distribution of MAA and B20. | One day prior to SIRT
  elimination half-life calculated in [min] from the decay-corrected radioactivity concentration measured over the liver; % radioactivity trapped in the liver at the individual measuring time points (of total radioactivity measured over the liver in the first scan); percent lung shunt (percentage of liver activity leaking to the lung at the individual time points)
Adverse events as elicited upon indirect questioning. | At any visit.
  Number of patients with adverse events (AEs), number of AEs per patient; descriptive listing of all AEs

CONTACTS AND LOCATIONS:
Overall Officials: Jens Ricke, Prof. Dr., Principal Investigator — University of Magdeburg, Faculty for Medicine
Locations (1):
- Clinic for Radiology and Nuclear Medicine, Magdeburg, Saxony-Anhalt, Germany